CLINICAL TRIAL: NCT05524129
Title: Evaluation of Adherence, Effect and Satisfaction With an Exercise Program in Patients With Chronic Low Back Pain - A Randomized Study
Brief Title: An Exercise Program in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ladislav Batalik, Principal Investigator, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vertebro-RHB_RHO/NK2022
Record Dates: First submitted 2022-08-23; First posted 2022-09-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Physiotherapy; Telerehabilitation
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Group I) (Experimental): It will be a hybrid form of rehabilitation, i.e. home exercises according to brochures in combination with regular visits to the ambulance for check-ups according to a precisely set schedule, the authorized physiotherapist will also contact the patients by phone at regular weekly intervals, thereby maintaining their motivation.
  Interventions: Other: rehabilitation exercise
- Control (Group II) (Active Comparator): These patients will undergo regular rehabilitation only in the outpatient center with the normally indicated frequency visits twice a week for 4 weeks.
  Interventions: Other: rehabilitation exercise; Other: electrotherapy

INTERVENTIONS:
Other: rehabilitation exercise — Conventional rehabilitation exercise.
Other: electrotherapy — A middle frequency electro-therapy
  Arms: Control (Group II)

SUMMARY:
Exercise intervention aims to improve the function of the deep back muscles and spine stabilizers, which appear to be an essential factor in preventing low back pain recurrences. In order to achieve the best possible effect of exercise, the patient should exercise for a long time even after finishing the exercise program, and it is also essential that exercises improve the function of the deep back muscles and become a regular part of the patient's life. In cooperation with the Neurological Clinic and physiotherapists from the Rehabilitation Department of the Brno University Hospital, the investigators put together a rehabilitation program to improve the function of the deep back muscles and spine stabilizers (group I). This program contains commonly used exercises; the patient can perform the exercises himself at home after the training, and no special aids are needed. The rehabilitation program is based on daily independent exercise, while the patient keeps a record of his activity in an exercise diary, which should contribute to motivation for regular exercise. At the same time, the physiotherapist will contact the patients by phone at regular weekly intervals, thereby maintaining their motivation. A total of 3 exercises were created, in which the patient will be taught gradually, according to his abilities and exercise tolerance. Regular checks with a physiotherapist are established to evaluate the correctness of the exercises, frequency, and effect and to increase the difficulty of the exercises. At the end of the exercise program, the patient will be instructed that it is desirable to continue the regular exercise. That exercise should become a part of everyday life to prevent the recurrence of vertebral disorders.

As part of our previous study entitled "Changes in the lumbar paraspinal muscles in patients with lower back pain," preliminary results showed a positive effect on the clinical condition of the patients, good tolerance of the exercises on the part of the patients, and satisfaction with completing the rehabilitation program.

DETAILED DESCRIPTION:
Patients with chronic lower back pain, eligible for study inclusion at the outpatient clinic of the Rehabilitation Department of the Brno University Hospital, will be randomized by an authorized physiotherapist into one of two groups. Interventional group, where a hybrid form of rehabilitation will be delivered. According to brochures, home-based exercises and regular outpatient visits will be delivered by a physiotherapist. Moreover, regular phone contact at weekly intervals will be provided for maintaining patient motivation. Control group, where patients will undergo regular rehabilitation-only in the outpatient center with the usually indicated frequency visits twice a week for 4 weeks).

In the experimental intervention, the exercise program is based on patient education, home-based individual training, and regular check-ups by a physiotherapist. The patients will also explain the importance of regular training and receive a booklet with photographed and described exercises. The patients will record their exercise frequency in a previously prepared diary - record sheet, which should also increase the patient's motivation to exercise. The first check-up with the physiotherapist will be 2 weeks from the start of the exercise to check the correct execution and regularity. The next check-up with the physiotherapist will be after 4 weeks, when the physiotherapist will recheck the current exercises. After the physiotherapist finds that the patient can perform individual exercises without problems, the difficulty of exercise will be increased (the patient receives another booklet with new, more challenging exercises). The same control and increase in the exercise's difficulty will occur after another 6 weeks. The total duration of the exercise program is 18 weeks.

In the control group, patients will be offered regular rehabilitation, including electrotherapy, and visits will be 2 times a week. The total duration of the rehabilitation program will be 4 weeks.

At the beginning and the end of the rehabilitation program, the disability of all patients will be evaluated using the Rolland-Morris questionnaire, the intensity of back pain, the quality of life using the short-form questionnaire, and the endurance of the trunk extensors (Biering-Sørensen test). At the end of the rehabilitation program, the patient will also evaluate his overall satisfaction with the completed rehabilitation program. The patient will be invited for a check-up 6 months after the end of the rehabilitation program to assess the same parameters that were assessed at the end of the program and to find out whether the patient continues to exercise regularly on his own.

Patients of both groups will undergo the exact measurements, which will then be statistically compared between the two groups.

The investigators plan to include 60 patients in the project.

ELIGIBILITY:
Inclusion Criteria:

* The cause of the problems most likely lies in the back area (e.g., dysfunction of trunk stabilization, faulty posture, inappropriate movement habits, beginning mild degenerative changes of the spine)
* age over 18 years (upper limit not determined)
* chronic lower back pain (pain duration of at least 12 weeks) - especially non-specific pain (pain localized in the lumbar spine or pain with propagation above the knee at the most), chronic radicular pain of vertebral etiology (not requiring rehabilitation aimed at paresis) can also be present.
* All patients enrolled in the study must have had an imaging examination of the lumbar spine.

Exclusion Criteria:

* overall poor physical condition, it should be noted that the patient must undergo entrance and exit examinations with a physiotherapist as part of the study, which requires a certain level of physical fitness
* involvement of the lumbar spine by another pathology (fracture, inflammation, tumor)
* the presence of comorbidity affecting the overall mobility of the patient (e.g., the presence of paresis after a stroke, severe heart failure leading to immobilization)
* significant impairment of cognitive functions (restricting cooperation in the study and filling out questionnaires)
* the patient is not motivated to exercise regularly to strengthen the paraspinal muscles
* back pain arose acutely (e.g., acute disc herniation, injury, acute blockage
* lower limb problems cause back pain (arthrosis, dysplasia, longer lower limb, one-sided flat feet) and problems with internal organs (inflammation of the bladder, kidneys, genitals)
* arthrosis of the hip, knee, and shoulder joints higher than grade II
* cachexia, obesity grade II to III,

Comment:

* the presence of milder chronic radiculopathy does not matter for entry into the study (muscle strength of lower limbs in individual segments should be at least IV grade)
* condition after lumbar spine surgery for degenerative changes in the anamnesis (more than 6 months) does not affect inclusion if the patient's condition allows exercise
* the exercise program can be adjusted individually according to the patient's condition
* it is necessary to have a signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline Functioning and disability score at 18 weeks and 6 months | Baseline, 18 weeks, 6 months
  Patient functioning and disability will be measured by the Roland-Morris Disability Questionnaire. Values ranges from 0-24, lower scores mean a better outcome.
Change from baseline Health-related quality of life score at 18 weeks and 6 months | Baseline, 18 weeks, 6 months
  Short Form Survey (SF-36) - 36-item. Maximum value is 100 points, minimum value is 36 point. Higher score mean a better outcome.
Change from baseline Endurance of the trunk extensors value at 18 weeks and 6 months | Baseline, 18 weeks, 6 months
  With the Biering-Sorensen Test, the patient's trunk extensors' endurance will be evaluated. Patients will be positioned in the prone position with the pelvis, hips, and knees in complete contact with the treatment bed. The patient's pelvis will be supported with a belt and fixed by the physiotherapist. The patients were asked to extend their upper body straight forward from the edge of the table and stay in this position. The time able to hold position properly will be recorded in seconds.

SECONDARY OUTCOMES:
Satisfaction - self-completed questionnaire | 18 week
  Patients will be provided with a 5-item self-completed questionnaire developed by our research team that will measure their satisfaction with the intervention they received and the study in general. The items will be presented in the form of statements to which patients will be asked to respond using a 1-5 Likert scale ("strongly agree", "agree", "not sure", "disagree", and strongly disagree").
Exercise adherence | 18 week
  Adherence to the exercise will be recorded in the data-sheets.The overall completion rate of prescribed exercise lessons in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Blanka Adamova, MD., PhD, Study Chair — Department of Neurology, University Hospital Brno, Czech Republic; Peter Krkoška, MD, Study Director — Department of Neurology, University Hospital Brno, Czech Republic; Filip Dosbaba, PT., PhD, Study Director — Department of Rehabilitation, University Hospital Brno, Czech Republic
Locations (1):
- Michaela Sládečková, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No